CLINICAL TRIAL: NCT06864923
Title: Investigation of the Effect of Hot Foot Bath on Sleep Quality and Fatigue
Brief Title: The Effect of Hot Foot Bath on Sleep Quality and Fatigue
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Uludag University (Other)
Responsible Party: Principal Investigator, Dilek Yilmaz, PhD, Associate Professor, Bursa Uludag University, Department of Nursing, Uludag University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2023-28/12
Record Dates: First submitted 2025-03-03; First posted 2025-03-07 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Hepatitis B
Keywords: fatigue; sleep quality; foot bath
MeSH Terms: conditions — Hepatitis B; Fatigue; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hot foot bath application group (Experimental)
  Interventions: Other: Hot foot bath application group
- Control group (No Intervention)

INTERVENTIONS:
Other: Hot foot bath application group — The intervention group will receive hot foot baths for three consecutive nights starting from the second day of hospitalization. The foot bath will be applied one hour before the patient goes to bed at night. The foot tub will be filled with hot water to approximately 20 cm above the patient's ankle and the temperature of the water will be measured with a water thermometer. The temperature of the water will be kept stable at 41-42°C. This application will be done for 20 minutes. The sleep and fatigue levels of the patients will be measured with measurement tools in the morning (3 times) following each application.
  Arms: Hot foot bath application group

SUMMARY:
This study will be conducted to investigate the effects of hot foot baths on patients' sleep quality and fatigue severity levels.The study will be conducted in the Gastroenterology clinic of a university hospital in Türkiye. The research sample will consist of 60 adult patients. Patients will be randomly divided into two groups: the intervention and control groups. The intervention group will receive hot foot baths for three consecutive nights starting from the second day of hospitalization. The foot bath will be applied one hour before the patient goes to bed at night. The foot tub will be filled with hot water to approximately 20 cm above the patient's ankle and the temperature of the water will be measured with a water thermometer. The temperature of the water will be kept stable at 41-42°C. This application will be done for 20 minutes. The sleep and fatigue levels of the patients will be measured with measurement tools in the morning (3 times) following each application. No application will be applied to the control group, and sleep and fatigue levels will be measured in a similar manner to the measurement tools applied to the intervention group and the application days.

ELIGIBILITY:
Inclusion Criteria:

* being over the age of 18,
* having no disorder which could affect pain perception,
* having no communication problem, and voluntarily agreeing to participate in the research,
* Having been admitted to the clinic at least 24 hours ago,
* Not having a diagnosed sleep disorder,
* Not having a psychiatric disorder requiring treatment,
* Not having a problem with vital signs before the application,
* Not using narcotic drugs in the last 4 hours,
* Not eating two hours before going to bed at night

Exclusion Criteria:

* being under the age of 18
* not being conscious, refusing to participate in the research or opting to leave the study at any point,
* Having a problem with vital signs before the application,
* Having a diagnosed sleep disorder.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-03-05 (Estimated); Primary Completion 2025-06-05 (Estimated); Study Completion 2025-06-05 (Estimated)

PRIMARY OUTCOMES:
fatigue severity in score (0-10) | 4 months
  Brief Fatigue Inventory: Scoring ranges from "0" to "10", with "0" indicating no effect and "10" indicating the highest level of effect. The general fatigue score is calculated by dividing the total score of items 1, 2 and 3 by 3, and the effect score of fatigue on daily living activities is calculated by dividing the total score of items 4a, 4b, 4c, 4d, 4e and 4f by 6. A score of "0" obtained from the KYE indicates no fatigue, "1-3" indicates low fatigue, "4-6" indicates moderate fatigue, "7-9" indicates high fatigue and "10" indicates the highest level of effe
Sleep Quality in score | 4 months
  Sleep Quality Scale: It consists of a total of 18 items. It includes items related to the sleep process and sleep satisfaction.

SECONDARY OUTCOMES:
weight | 4 months
  weight in kilograms

IPD SHARING:
Plan to Share IPD: Undecided